CLINICAL TRIAL: NCT03303118
Title: The Effects of Hypobaria vs Hypoxia on Cerebral Vasoreactivity, Brain's Electrical Activity and Concentration Performance on Pilots.
Brief Title: The Effects of Hypobaria vs Hypoxia on Cerebral Functions.
Acronym: Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fliegerärztliches Institut (Other)
Responsible Party: Principal Investigator, Mathias Aebi, PhD, Dr. med Denis Bron, Fliegerärztliches Institut
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-00752
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Cerebral Hypoxia
Keywords: Hypoxia; Brain; Cerebral vaso-reactivity; EEG; Concentration performance; Cerebral oxygenation; Cerebral blood-flow; Heart rate variability
MeSH Terms: conditions — Hypoxia, Brain; Hypoxia

STUDY DESIGN:
Intervention Model Description: Single-Blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Left (Other): No product administration will be done in this study.
  Interventions: Other: Hypoxia

INTERVENTIONS:
Other: Hypoxia — No drug or product will be used in this study. No medication will be give to the participants. No arm will be used for product administration.

SUMMARY:
The investigators will investigate the effect of hypobaria and hypoxia on physiological responses such as: oxygen saturation, heart rate, cerebral blood flow, cerebral oxygenation, brain's activity and concentration performance.

DETAILED DESCRIPTION:
The main goal of this project is to investigate how hypoxia affects cognitive functions. The KLT-R test asses the concentration level of a person. Subjects will do this test at different simulated altitude level in the hypobaric chamber at the FAI in Dübendorf. Investigators' first hypothesis is that concentration level will be altered by hypoxia. The higher altitude the subjects are, the more the concentration would be altered. KLT-R performance would be impaired by hypoxia compare to sea level performance.

The primary endpoint of this project is to investigate how KLT-R performance is affected by the different hypoxic conditions. KLT-R test will be passed nine times in total during the test visit. There will be a pre-test; a test at each of the conditions (3000m HH, 5500m HH, 5500m NH and 5500m HN); between each condition at sea level (to have a new baseline before each condition) and a post-test at the end of the protocol. To avoid influence of fatigue, all conditions will be randomized.

The second endpoint of this study is how the brain electrical activity is modulated by hypoxia. Micro-states also will be measure during hypobaric hypoxia conditions (3000m HH and 5500m HH).

ELIGIBILITY:
Inclusion Criteria:

* No history of flight sickness
* No relevant medical diseases
* Age 18 - 40 years
* Written consent acceptance

Exclusion Criteria:

* Known pathologies
* Relevant medical disorders
* Drug addiction
* Anemia or poor health
* People who have already had problems with elevation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Concentration performance | 4 minutes per test
  Performance of concentration at different altitude levels.

SECONDARY OUTCOMES:
EEG micro-states | 5 minutes per record
  5 minutes recording in each conditions, eyes closed, at rest.

OTHER OUTCOMES:
Cerebral vaso-reactivity | 8 Minutes per test
  Cerebral vasoreactivity after 1 minute hyperventilation and 3 minutes breathing of 5% CO2 mixture.

CONTACTS AND LOCATIONS:
Locations (1):
- Mathias Aebi, Dübendorf, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Results will be shared in scientific publications by the end of this year and in 2018.

REFERENCES:
- [Derived] Aebi MR, Bourdillon N, Kunz A, Bron D, Millet GP. Specific effect of hypobaria on cerebrovascular hypercapnic responses in hypoxia. Physiol Rep. 2020 Feb;8(4):e14372. doi: 10.14814/phy2.14372. PMID 32097541